CLINICAL TRIAL: NCT07348029
Title: Investigation of the Distance of the Needle Entry Point From the Anus and the Depth to Reach the Pudendal Nerve in Pudendal Nerve Block Application in Children
Brief Title: Anatomical Measurements of Pudendal Nerve Block in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Münevver Kayhan, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: ctf- pudental mesafe- 04
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management; Penile Surgery-Related Pain
Keywords: Pudendal Nerve Block; Pediatric Regional Anesthesia; Neurostimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Penile Surgery Cohort: Children aged 1-18 years undergoing penile surgery with neurostimulation-guided pudendal nerve block; anatomical measurements of needle insertion distance from anus and nerve depth are recorded.
  Interventions: Procedure: Neurostimulation-Guided Pudendal Nerve Block

INTERVENTIONS:
Procedure: Neurostimulation-Guided Pudendal Nerve Block — Bilateral pudendal nerve block is performed under general anesthesia with neurostimulation guidance. Anatomical measurements, including distance from anus to needle insertion point and nerve depth, are recorded for each patient. Bupivacaine 0.25% is used at 0.25 ml/kg per side, with a maximum total dose of 2 mg/kg.

SUMMARY:
This prospective observational study aims to investigate the relationship between anatomical parameters-specifically the distance from the anus to the needle insertion point and the depth required to reach the pudendal nerve-during neurostimulation-guided pudendal nerve block and patients' age, height, and weight in children undergoing penile surgery.

DETAILED DESCRIPTION:
The pudendal nerve originates from the sacral nerve roots Sacral2-Sacral4 and provides sensory and motor innervation to the penile and perineal regions. Effective postoperative analgesia is essential in pediatric penile surgeries. Pudendal nerve block may provide longer-lasting and more effective analgesia compared to caudal or penile blocks.

However, due to age- and size-related anatomical variability in children, data regarding optimal needle insertion distance and depth to reach the pudendal nerve are limited. In this study, neurostimulation will be used to confirm pudendal nerve localization, and anatomical measurements will be analyzed in relation to demographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years
* Scheduled for penile surgery (e.g., hypospadias, phimosis)
* Planned to receive neurostimulation-guided pudendal nerve block
* Patient and parents/legal guardians willing to participate under general anesthesia

Exclusion Criteria:

* Patients with incomplete measurement data
* Cases where successful nerve block cannot be performed or nerve stimulation is not detectable at currents ≥1.5 mA
* Patients or parents/legal guardians who refuse pudendal nerve block
* Patients with pelvic deformities or neuromuscular disorders

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study includes children aged 1-18 years who are undergoing penile surgery. Neurostimulation-guided pudendal nerve block will be performed, and anatomical measurements, including the horizontal distance from the anus to the needle insertion point and the depth from the skin to the pudendal nerve, will be recorded. Measurements will be taken separately for the right and left sides. Patient age, height, and weight will also be recorded, and their relationship with the anatomical measurements will be analyzed. The study will be conducted at Istanbul University-Cerrahpasa, Department of Pediatric Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Horizontal distance from anus to needle insertion point and Depth from skin surface to pudendal nerve | During pudendal nerve block procedure
  The horizontal distance from the anus to the needle insertion point is measured in centimeters for each patient using neurostimulation-guided pudendal nerve block. Measurements are recorded separately for the right and left sides.The depth from the skin surface to the pudendal nerve is measured in centimeters using neurostimulation guidance. Measurements are recorded separately for the right and left sides. The relationship of this distance and the association of nerve depth with patient age, height, and weight will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Munevver Kayhan, Lecturer Doctor, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Pinar Kendigelen, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Ayse Cigdem Tutuncu, Professor Doctor, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty, Bakırköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015
- [Result] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928